CLINICAL TRIAL: NCT03266861
Title: Study of Transcutaneous Exercise Oxymetry, reLationship to LActates Increase in Claudication
Brief Title: Lactate Increase in Peripheral Artery Disease
Acronym: STELLA
Status: Completed | Type: Observational
Sponsor: University Hospital, Angers (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2017-A00912-51
Record Dates: First submitted 2017-08-22; First posted 2017-08-30 (Actual); Last update posted 2021-07-12 (Actual); Status verified 2020-08

CONDITIONS: Peripheral Artery Disease; Claudication, Intermittent
MeSH Terms: conditions — Peripheral Arterial Disease; Intermittent Claudication

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients undergoing exercise oximetry: Patients with PAD referred for treadmill testing and exercise oximetry
  Interventions: Diagnostic Test: Exercise oximetry

INTERVENTIONS:
Diagnostic Test: Exercise oximetry — Sample at rest before the walking test Sample at rest 3 minutes after the end of the walking period
  Other Names: Capillary blood sampling from the earlobe

SUMMARY:
To our knowledge, the measurement of the transcutaneous oxygen pressure during walking is the only continuous method that estimates the importance of ischemia, bilaterally and segment of limb by segment of limb. The determination of the lactates concentration, with micro method from earlobe sampling, is very widely validated in physiology and exercise physiopathology; and it is widely used, by laboratories, for exercise investigation in athletes. We use it in routine to evaluate the presence of functional limitation during tcpO2 tests on a treadmill.

The present study hypothesises a significant relationship between lactatemia variation (difference between lactatemia after 3 minutes of recovery from walking and the value at rest) and tcpO2 "decrease from rest of oxygen pressure (DROP) values for patients with peripheral artery disease (PAD).

DETAILED DESCRIPTION:
Lactates sample (100 microliter) will be collected at rest Ankle brachial index is measured at rest transcutaneous oxygen pressure is measured at the chest, calves and buttocks and results will be expressed as the minimal value of the DROP index (Limb changes minus chest changes) Patients walk on treadmill (2MPH 10% slope) until exertional limb pain. Lactates sample (100 microliter) will be collected at minute 3 of recovery from walking Correlation of lactate increase to the sum of DROP values wil be studied

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years old
* Patient able to walk on a treadmill
* Patient covered by the French health insurance
* Patient able to understand the protocol
* Patient agrees to be involve in the protocol and sign the consent form

Exclusion Criteria:

* Patient refuses to participate at the this protocol
* Patient has a wash-out period for another clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient with peripheral artery disease
Sampling Method: Non-Probability Sample
Enrollment: 750 (Actual)
Dates: Start 2017-10-03 (Actual); Primary Completion 2020-10-10 (Actual); Study Completion 2020-10-10 (Actual)

PRIMARY OUTCOMES:
Correlation of lactate results to oximetry | one and a half hour
  Evaluate the coefficient of correlation between the lactatemia increase from rest and the sum of the observed DROP values of all studied subjects.

SECONDARY OUTCOMES:
Correlation of lactate results to resting Ankle to brachial index (ABI) | one and a half hour
  Evaluate the coefficient of correlation between the lactatemia increase from rest and the sum of the resting ABI value of all studied subjects..

CONTACTS AND LOCATIONS:
Overall Officials: Pierre ABRAHAM, MD; PhD, Principal Investigator — University Hospitaml in Angers
Locations (1):
- Centre hospitalier universitaire, Angers, France

IPD SHARING:
Plan to Share IPD: Undecided